CLINICAL TRIAL: NCT06579378
Title: Virtual Sail 3D - A Feasibility Study for Enhancing Cognitive Functions in Elderly People
Brief Title: Feasibility Study of Virtual Sail 3D in Cognitive Functions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Collaborators: Fondazione di Sardegna (Unknown)
Responsible Party: Principal Investigator, Federica Sancassiani, Principal Investigator, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NP/2023/2557
Record Dates: First submitted 2024-08-21; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Virtual reality; Feasibility; Cognitive functions; Sail; Advances Technologies Laboratory
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VSail 3D (Experimental): The "VSail 3D" experimental protocol includes 12 sessions (2 times a week, for 6 consecutive weeks) with scenarios (virtual environments) dedicated to the sport of sailing.
  The duration of each session is 50-60 minutes.
  Interventions: Device: VSail 3D
- WEB-Health (Active Comparator): The intervention regards education on healthy lifestyles to promote active ageing (topics: physical activity in old age; effective communication, stress management, technologies and health). It will consist of 3 seminars, delivered in the form of webinars, on a bi-weekly basis over 6 consecutive weeks, lasting 50-60 minutes each.
  Interventions: Other: WEB-Health

INTERVENTIONS:
Device: VSail 3D — The "CEREBRUM" software with virtual sailing scenarios is made up of exercises of variable difficulty, designed to train different cognitive functions, in particular attention, memory, learning, cognitive estimates, working memory, executive functions, motor abilities and language. The different degrees of difficulty are designed to adapt to the user's functional diagnosis. The operator who conducts the intervention must adapt the difficulty level to the user's residual abilities, so that the exercises are neither too easy nor too complex. Each session, after an initial part of welcome, psychoeducation and orientation to the instrument, involves alternating virtual reality exercises, positive and corrective feedback, and suggestions of practical homework related to the cognitive function trained during the session that the individual should try during daily life.
  Arms: VSail 3D
Other: WEB-Health — The intervention includes a series of 3 webinars focused on active ageing promotion. In particular, each webinar will regard topics related to healthy lifestyle, such as physical activity in old age, effective communication, stress management, technologies and health. Each webinar will be conducted by a mental health professional, and it will be delivered in real-time in a group (plenary).
  Arms: WEB-Health

SUMMARY:
This research project will assess the feasibility and preliminary effectiveness of a 6-week intervention to improve cognitive functions using the 3D immersive virtual reality software "CEREBRUM" with virtual sailing scenarios among elderly with mild cognitive impairment. CEREBRUM, developed by PRoMIND in association with IDEGO, is the first European tool for enhancing cognitive functions via 3D immersive virtual reality in psychosocial disabilities. Previous studies have shown its effectiveness in improving cognitive functions and well-being in people with bipolar disorders. The software includes modules for memory, learning, cognitive estimations, attention, working memory, and executive functions. For this study, the software was developed with sailing virtual scenarios to make it more enjoyable and engaging, as well as to train other cognitive functions such as motor skills and language abilities among people with disabilities.

DETAILED DESCRIPTION:
Research on active aging has been identified as a priority, particularly concerning the feasibility and effectiveness of non-pharmacological interventions aimed at preventing and/or delaying cognitive decline. Risk factors such as physical, cognitive, and social inactivity are estimated to account for about 40% of the risk of developing dementia in the lifetime. Recent reviews have shown that cognitive remediation interventions are effective in improving cognitive performance in older adults with and without cognitive decline.

Cognitive remediation is a behavior-based training intervention aimed at improving cognitive functions (memory, attention, executive functions, social cognition, and metacognition) to achieve lasting results and their generalization. There is substantial evidence supporting the effectiveness of such interventions in neuropsychological disorders such as dementia, mild cognitive impairment, and behavioral disorders.

In recent years, there has been an increase in the use of immersive 3D virtual reality software in clinical and rehabilitative settings as tools for rehabilitation and the improvement of various skills. To date, there are few studies where immersive 3D virtual reality is used to enhance cognitive functions related to personal and social functioning, especially to prevent cognitive decline in older adults (aged 65 and over).

This research project will assess the feasibility and preliminary effectiveness of a 6-week intervention to improve cognitive functions using the 3D immersive virtual reality software "CEREBRUM" with sailing scenarious among elderly with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65 years or older
* Sex: all
* Living independently,
* Without conditions that would prevent them from participating in the activities of the experimental intervention "VSail 3D,"
* Without severe issues with autonomous mobility
* With Mild Cognitive Impairment (MCI) according to Addenbrooke's Cognitive Examination for cognitive functions (ACE-R), which also includes the Mini-Mental State Examination (MMSE), with the following ranges: ACE = 66.93-79.86 and/or MMSE = 21-25.
* Signing the informed consent

Exclusion Criteria:

* severe cardiovascular conditions
* severe issues with autonomous mobility
* severe metabolic disorders not pharmacologically compensated
* severe neurological conditions that prevent from participating in the experimental protocol, such as a stroke within the past 2 years, Parkinson's disease, epilepsy, or dementia (Alzheimer's, vascular, etc.)
* severe ongoing bronchopulmonary disorders
* severe ongoing renal disorders
* glaucoma, retinal detachment, or other serious vision conditions that do not allow the safe use of 3D virtual reality technology
* active malignant neoplasm that do not allow the hinders participation in the intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dropout rates; Proportion of recruited participants among those considered eligible; | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Feasibility will be assessed based on tolerability, including dropout rates and acceptability, which considers the proportion of recruited participants among those considered eligible.
Simulator Sickness Questionnaire (SSQ) | T0 (0 weeks) - T1 (6 weeks)
  Feasibility will be assessed based on side effects through the Simulator Sickness Questionnaire (SSQ), a self-report questionnaire that evaluates the frequency of unwanted effects that may occur due to the use of virtual reality technologies, such as nausea, dizziness, headaches, eye strain, etc. 16 items.
  The score range is 0-48, with higher scores indicating worse side effects.
Self-report satisfaction questionnaire | T1 (6 weeks)
  Feasibility will be assessed based on a Self-report satisfaction questionnaire, constructed ad hoc to evaluate the level of satisfaction with the program as a whole, the effect on psychophysical health, helping and listening abilities demonstrated by the operators, organizational support for activities, satisfaction with initial expectations.
  The score range is 6-30, with higher scores indicating higher satisfaction.

SECONDARY OUTCOMES:
Trail Making Test | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on executive functions
Digit Span | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on memory
Stroop Test | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on executive functions
Rey Figure Test | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on visual spatial function
Frontal Assessment Battery (FAB) | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on executive functions
Matrix test | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on selective attention
Rey's Word Test | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on memory
Addenbrooke's Cognitive Examination (ACE-R) | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on general cognitive functions, the neuropsychological tests is used to identify cognitive impairment in conditions such as dementia.

OTHER OUTCOMES:
Short Form Health Survey, 12 items (SF-12) | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on quality of life, 12 item. The score range il 12-47, with higher scores indicating better quality of life.
Patient Health Questionnaire (PHQ-9) | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on depressive symptoms, 9 Item. The score range is 0-27, with higher scores indicating worse depressive symptoms.
Generalized Anxiety Disorder-7 item (GAD-7) | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on anxiety, 7 item. The score range is 0-21, with higher scores indicating worse anxious symptoms.
Brief Social Rhythms Scale (BSRS) | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on dysregulation of biological and social rhythms, 10 item.
  The score range is 10-60, with higher scores indicating worse dysregulation of rhythms.
Physical Body Experiences Questionnaire Simplified for Active Aging (PBE-QAG) | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on body awareness in people over 65 years old, 12 item.
  The score range is 12-60, with higher scores indicating worse body awareness.
International Physical Activity Questionnaire (IPAQ) | T0 (0 weeks); T1 (6 weeks); T2 (12 weeks from T1); T3 (24 weeks from T1); T4 (36 weeks from T1); T5 (48 weeks from T1)
  Preliminary measure of effectiveness on level of physical activity carried out in the last 7 days, 9 item.
  The total score is based on the conventional unit of measure "MET," where higher MET correspond to higher levels of physical activity. Typically, a score of less than 700 MET indicates a low level of physical activity, a score between 700 and 2519 MET indicates a moderate level of physical activity, and a score greater than or equal to 2520 MET indicates an intense level of physical activity.
Sway area in the presence and absence of visual input | T0 (0 weeks); T1 (6 weeks)
  95% confidence ellipse calculated based on the center of pressure time-series acquired using a pressure baropodometric platform.
Gait speed | T0 (0 weeks); T1 (6 weeks)
  Speed calculated on a 20 m straight trajectory. This is obtained by processing the trunk accelerations recorded by a single wearable inertial sensor (BTS-G-Sensor2) located in the low back (L5-S1 vertebrae).
Timed up and go time | T0 (0 weeks); T1 (6 weeks)
  time needed to complete a 3m Timed-up-and-go (TUG) test. This will be carried out using a single wearable inertial sensor located in the low back (L2 vertebrae).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cagliari, Cagliari, CA, Italy

REFERENCES:
- [Derived] Sancassiani F, Perra A, Vacca V, Montisci R, Monni M, Lorrai S, Cossu G, Petretto DR, di Natale L, Primavera D, Redolfi S, Scuteri A, Nardi AE, Kalcev G, Pau M, Carta MG. Enhancing Cognitive Functions in Older Adults With Mild Cognitive Impairment via Virtual Sail 3D: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2026 Jan 15;15:e85089. doi: 10.2196/85089. PMID 41538788